CLINICAL TRIAL: NCT01195662
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 3 Trial to Evaluate the Safety and Efficacy of Dapagliflozin in Subjects With Type 2 Diabetes With Inadequately Controlled Hypertension on an Angiotensin-Converting Enzyme (ACE) Inhibitor or Angiotensin Receptor Blocker (ARB) and an Additional Antihypertensive Medication
Brief Title: A Study of BMS-512148 (Dapagliflozin) in Patients With Type 2 Diabetes With Inadequately Controlled Hypertension on an ACEI or ARB and an Additional Antihypertensive Medication
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB102-077 ST; 2010-019798-13 (EudraCT Number)
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Mellitus, Type 2; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases; Angiotensin Receptor Inhibitors; Angiotensin-Converting Enzyme Inhibitors; Antihypertensive Agents; Cardiovascular Agents; Pharmacological Actions
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin 10 mg (Experimental): Dapagliflozin 10 mg tablets
  Interventions: Drug: Dapagliflozin
- Placebo matching Dapagliflozin (Placebo Comparator): Placebo tablets matching dapagliflozin tablets
  Interventions: Drug: Placebo matching Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 10 mg, once daily, Up to 12 weeks
  Other Names: BMS-512148; Farxiga™
  Arms: Dapagliflozin 10 mg
Drug: Placebo matching Dapagliflozin — Tablets, Oral, 0 mg, once daily, Up to 12 weeks
  Arms: Placebo matching Dapagliflozin

SUMMARY:
The purpose of this study is to learn if BMS-512148 (Dapagliflozin), after 12 weeks, can improve (decrease) blood pressure in patients with type 2 diabetes with uncontrolled hypertension who are on an Angiotensin-converting enzyme inhibitor (ACEI) or an Angiotensin Receptor Blocker (ARB).The safety of this treatment will also be studied

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Males and females, 18 to 89 years old, with type 2 diabetes with inadequate glycemic control HbA1c between 7-10.5% and uncontrolled hypertension Systolic Blood Pressure (SBP) 140-165 and Diastolic Blood Pressure (DBP) 85-105
* Subjects must have a mean 24 hr blood pressure ≥ 130/80 determined by Ambulatory Blood Pressure Monitoring (ABPM) within 1 week prior to Day 1 visit
* Stable dose of oral antidiabetic agent (OAD) for at least 6 weeks [12 wks for Thiazolidinedione (TZD)] or a stable daily dose of insulin, as a monotherapy or in combination with another OAD, for 8 weeks, and a stable dose of ACEI or ARB and 1 additional antihypertensive medication for at least 4 weeks
* C-peptide ≥ 0.8 ng/mL
* Body Mass Index ≤ 45.0 kg/m2
* Serum creatinine < 1.50 mg/dL for men or < 1.40 mg/dL for women

Exclusion Criteria:

* Aspartate aminotransferase (AST) and /or Alanine aminotransferase (ALT) > 3.0*upper limit of normal (ULN)
* Serum total bilirubin ≥ 1.5*ULN
* Creatinine kinase > 3*ULN
* Symptoms of severely uncontrolled diabetes
* History of malignant or accelerated hypertension
* Currently unstable or serious cardiovascular, renal, hepatic, hematological, oncological, endocrine, psychiatric, or rheumatic diseases

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2245 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (274):
- United States (155):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Wilmax Clinical Research, Inc., Mobile, Alabama
  - 43rd Medical Associates, Phoenix, Arizona
  - Central Phoenix Medical Center, Tempe, Arizona
  - Clinical Research Advantage, Inc./Mesa Family Med Ctr, Pc, Tempe, Arizona
  - Clinical Research Advantage/Desert Clinical Research, Tempe, Arizona
  - Visions Clinical Research - Tucson, Tucson, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Aureus Research, Inc., Little Rock, Arkansas
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Cmp Research, Anaheim, California
  - Catalina Research Institute, Llc, Chino, California
  - Southland Clinical Research Center, Inc., Fountain Valley, California
  - Marin Endocrine Care & Research, Inc., Greenbrae, California
  - Del Rosario Medical Clinic, Inc., Huntington Park, California
  - Time Clinical Research Inc., Huntington Park, California
  - Clinica Medica San Miguel, Los Angeles, California
  - American Institute Of Research, Los Angeles, California
  - Randall G. Shue, D.O., Los Angeles, California
  - Mcs Clinical Trials, Los Angeles, California
  - National Research Inst, Los Angeles, California
  - Diabetes Medical Center Of California, Northridge, California
  - Valley Clinical Trials, Northridge, California
  - Lucita M. Cruz,Md.,Inc., Norwalk, California
  - Sds Clinical Trials, Orange, California
  - Bayview Research Group, Llc, Paramount, California
  - San Diego Managed Care Group, Poway, California
  - Integrated Research Group, Inc., Riverside, California
  - Quality Control Research, Inc, Sacramento, California
  - Wetlin Research Associates, Inc., San Diego, California
  - Crest Clinical Trials, Inc., Santa Ana, California
  - Neurological Research Institute, Santa Monica, California
  - Orrin M. Troum, Md And Medical Associates, Santa Monica, California
  - Torrance Clinical Research, Torrance, California
  - Orange County Research Center, Tustin, California
  - University Clinical Investigators, Inc., Tustin, California
  - Chase Medical Research, Llc, Waterbury, Connecticut
  - Christiana Care Health Services, Inc, Newark, Delaware
  - Zasa Clinical Research, Boynton Beach, Florida
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Innovative Research Of West Florida, Inc, Clearwater, Florida
  - Clinical Research Of South Florida, Coral Gables, Florida
  - Avail Clinical Research, Llc, DeLand, Florida
  - International Research Associates, Llc, Hialeah, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - The Community Research Of South Florida, Hialeah, Florida
  - Central Florida Internists, Kissimmee, Florida
  - Flcri Global Research, Llc, Miami, Florida
  - Clinical Research Of Miami, Inc., Miami, Florida
  - Pharmax Research Clinic, Inc., Miami, Florida
  - Apf Research, Llc, Miami, Florida
  - Community Research Foundation, Inc., Miami, Florida
  - Baptist Diabetes Associates, Pa, Miami, Florida
  - Newphase Clinical Trials, Inc., Miami Beach, Florida
  - Ocean Blue Medical Research Center, Inc., Miami Springs, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Florida Institute For Clinical Research, Llc, Orlando, Florida
  - Michele A. Morrison Internal Medicine, Inc., Pembroke Pines, Florida
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - Meridien Research, Tampa, Florida
  - Perimeter Institute For Clinical Research, Atlanta, Georgia
  - Bainbridge Medical Associates, Bainbridge, Georgia
  - River Birch Research Alliance, Llc, Blue Ridge, Georgia
  - In-Quest Medical Research, Llc, Duluth, Georgia
  - Middle Georgia Drug Study Center, Llc, Perry, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - So. Illinois Clin Res Ctr @ Div Of Kevin L Pritchett Md, Pc, O'Fallon, Illinois
  - Springfield Diabetes And Endocrine Center, Springfield, Illinois
  - American Health Network Of Indiana Llc, Avon, Indiana
  - Investigators Research Group, Llc, Brownsburg, Indiana
  - American Health Network Of In Llc, Franklin, Indiana
  - Laporte County Institute For Clinical Research, Inc., Michigan City, Indiana
  - American Health Network Of In Llc, Muncie, Indiana
  - Medical Development Centers, Llc, Baton Rouge, Louisiana
  - Omega Clinical Research, Llc, Metairie, Louisiana
  - Acadia Clinical Research, Llc, Bangor, Maine
  - Alternative Primary Care, Silver Spring, Maryland
  - Hci-Metromedic Walk-In Medical Office, New Bedford, Massachusetts
  - Neurocare, Inc., Newton, Massachusetts
  - Atlantic Clinical Trials, Llc, Watertown, Massachusetts
  - Providence Park Clinical Research, Novi, Michigan
  - The Center For Clinical Trials, Biloxi, Mississippi
  - Phillips Medical Services, Pllc, Jackson, Mississippi
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Kcumb Dybedal Clinical Research Center, Kansas City, Missouri
  - Clin Research Advantage, Inc. James Meli, Do Family Pracice, Henderson, Nevada
  - Office Of Ted Thorp, Md, Las Vegas, Nevada
  - Independent Clinical Researchers@ Wolfson Medical Center, Las Vegas, Nevada
  - Clinical Research Advantage, Inc., Las Vegas, Nevada
  - Palm Medical Research Center, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Premier Research, Trenton, New Jersey
  - Medex Healthcare Research, Inc., New York, New York
  - Digiovanna Institute For Medical Education & Research, North Massapequa, New York
  - Southgate Medical Group, West Seneca, New York
  - Diabetes & Endocrinology Consultants, Morehead City, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Community Health Care, Inc., Canal Fulton, Ohio
  - Community Research, Cincinnati, Ohio
  - Parsons Avenue Medical Clinical, Columbus, Ohio
  - Clinical Research Source, Inc, Perrysburg, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Integris Family Care Yukon, Yukon, Oklahoma
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - Southeastern Pa Medical Institute, Broomall, Pennsylvania
  - Abington Memorial Hos/Feasterville Family Health Care Center, Feasterville, Pennsylvania
  - The Clinical Trial Center, Llc, Jenkintown, Pennsylvania
  - Arcuri Clinical Research Llc, Philadelphia, Pennsylvania
  - Philadelphia Health Associates - Adult Medicine, Philadelphia, Pennsylvania
  - Research Across America, Reading, Pennsylvania
  - Pish Medical Associates, Uniontown, Pennsylvania
  - Greater Providence Clinical Research, Llc, Warwick, Rhode Island
  - Medical Research South, Charleston, South Carolina
  - Southeastern Research Associates, Inc., Greenville, South Carolina
  - North Myrtle Beach Family Practice, North Myrtle Beach, South Carolina
  - Pawleys Pediatrics And Adult Medicine, Pawleys Island, South Carolina
  - Hillcrest Clinical Reseach, Llc, Simpsonville, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Southwind Medical Specialists, Memphis, Tennessee
  - Tn Medical Research, Spring Hill, Tennessee
  - Arlington Family Research Center, Inc., Arlington, Texas
  - 3rd Coast Research Associates, Corpus Christi, Texas
  - Krk Medical Research, Dallas, Texas
  - Research Institute Of Dallas, Dallas, Texas
  - Internal Medicine Clinical Reaseach, Dallas, Texas
  - Renaissance Clinical Research And Hypertension Pllc, Dallas, Texas
  - Sergio F. Rovner, M.D., El Paso, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Village Family Practice, Houston, Texas
  - Dependable Clinical Research, Llc, Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Bellaire Medical Care Group, Houston, Texas
  - Excel Clinical Research, Llc, Houston, Texas
  - Hill Country Medical Associates, New Braunfels, Texas
  - North Hills Medical Research, Inc., North Richland Hills, Texas
  - Med-Olam Clinical Research, Pasadena, Texas
  - Lisa E. Medwedeff, Md, Pa, Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Abbott Clinical Research Group, Inc., San Antonio, Texas
  - Covenant Clinical Research, Pa, San Antonio, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Breco Research, Ltd, Sugarland, Texas
  - Exodus Healthcare Network, Magna, Utah
  - Wasatch Endocrinology And Diabetes Specialists, Salt Lake City, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Alexandria Health Care Center, Alexandria, Virginia
  - Millennium Clinical Trials Llc, Arlington, Virginia
  - Burke Internal Medicine And Research, Burke, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Hampton Roads Center For Clinical Research, Inc., Suffolk, Virginia
  - Larry D. Stonesifer, Md, Federal Way, Washington
  - Sound Medical Research, Port Orchard, Washington
  - Clinical Investigation Specialists, Inc., Kenosha, Wisconsin
- Australia (3):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Nedlands, Western Australia
- Canada (7):
  - Local Institution, Kelowona, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Monction, New Brunswick
  - Local Institution, Brampton, Ontario
  - Local Institution, Granby, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Colombia (4):
  - Local Institution, Armenia, Quindío Department
  - Local Institution, Bucaramanga, Santander Department
  - Local Institution, Barranquilla
  - Local Institution, Bogotá
- Czechia (7):
  - Local Institution, Beroun
  - Local Institution, Cheb
  - Local Institution, Havířov
  - Local Institution, Krnov
  - Local Institution, Liberec
  - Local Institution, Ostrava
  - Local Institution, Prague
- Denmark (4):
  - Local Institution, Copenhagen
  - Local Institution, Frederiksberg
  - Local Institution, Gentofte Municipality
  - Local Institution, Slagelse
- Finland (4):
  - Local Institution, Helsinki
  - Local Institution, Kerava
  - Local Institution, Kokkola
  - Local Institution, Oulu
- Germany (17):
  - Local Institution, Aschaffenburg, Bavaria
  - Local Institution, Augsburg, Bavaria
  - Local Institution, Duisburg, North Rhine-Westphalia
  - Local Institution, Bad Kreuznach
  - Local Institution, Berlin
  - Local Institution, Dortmund
  - Local Institution, Dresden
  - Local Institution, Karlsruhe
  - Local Institution, Köthen
  - Local Institution, Kronshagen
  - Local Institution, Langenfeld
  - Local Institution, Lüneburg
  - Local Institution, Magdeburg
  - Local Institution, Mainz
  - Local Institution, Mannheim
  - Local Institution, Saarbrücken
  - Local Institution, Wüstensachsen
- Hungary (10):
  - Local Institution, Gyöngyös, Heves County
  - Local Institution, Budapest
  - Local Institution, Eger
  - Local Institution, Kisvárda
  - Local Institution, Miskolc
  - Local Institution, Nyíregyháza
  - Local Institution, Sátoraljaújhely
  - Local Institution, Sopron
  - Local Institution, Szeged
  - Local Institution, Szekszárd
- India (15):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Mangalore, Karnataka
  - Local Institution, Belagavi, Karnatka
  - Local Institution, Indore, Madhya Pradesh
  - Local Institution, Nagpur, Maharashtra
  - Local Institution, Delhi, New Delhi
  - Local Institution, Jaipur, Rajasthan
  - Local Institution, Chennai, Tamil Nadu
  - Local Institution, Coimbatore, Tamil Nadu
  - Local Institution, Madurai, Tamil Nadu
  - Local Institution, Chennai Tamilnadu
  - Local Institution, Hyderabad
  - Local Institution, Nagpur
  - Local Institution, Trivandrum
- Ireland (2):
  - Local Institution, Dublin, Dublin
  - Local Institution, Galway
- Mexico (12):
  - Local Institution, Chihuahua City, Chihuahua
  - Local Institution, Torreón, Coahuila
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Distrito Federal, Mexico City
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Tlalpan, Mexico City
  - Local Institution, Cuautla, Morelos
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, San Luis Potosí City, San Luis Potosí
  - Local Institution, Culiacán, Sinaloa
  - Local Institution, Mérida, Yucatán
  - Local Institution, Del. Benito Juarez
- Poland (16):
  - Local Institution, Gdynia, Gdynia
  - Local Institution, Bialystok
  - Local Institution, Chrzanów
  - Local Institution, Elblag
  - Local Institution, Gdansk
  - Local Institution, Kamieniec Ząbkowicki
  - Local Institution, Katowice
  - Local Institution, Kielce
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Lublin
  - Local Institution, Ostróda
  - Local Institution, Poznan
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
  - Local Institution, Zabrze
- Puerto Rico (3):
  - Local Institution, Fajard
  - Local Institution, Ponce
  - Local Institution, San Juan
- Romania (11):
  - Local Institution, Oradea, Bihor County
  - Local Institution, Oradea, Jud. Bihor
  - Local Institution, Timișoara, Jud. Timis
  - Local Institution, Târgu Mureş, Mureș County
  - Local Institution, Ploieşti, Prahova
  - Local Institution, Satu Mare, Satu Mare County
  - Local Institution, Sibiu, Sibiu County
  - Local Institution, Timișoara, Timiș County
  - Local Institution, Bucharest
  - Local Institution, Cluj-Napoca
  - Local Institution, Sibiu
- United Kingdom (4):
  - Local Institution, Irvine, Ayrshire
  - Local Institution, Ely, Cambridgeshire
  - Local Institution, Birmingham, West Midlands
  - Local Institution, Bath, Wiltshire

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Weber MA, Mansfield TA, Cain VA, Iqbal N, Parikh S, Ptaszynska A. Blood pressure and glycaemic effects of dapagliflozin versus placebo in patients with type 2 diabetes on combination antihypertensive therapy: a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Diabetes Endocrinol. 2016 Mar;4(3):211-220. doi: 10.1016/S2213-8587(15)00417-9. Epub 2015 Nov 27. PMID 26620248
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment: 29-Oct-2010 to 04-Oct-2012. Original study had 3 arms but 5 mg dapagliflozin arm was discontinued with Protocol Amendment 8 (implemented 01-Nov-2011) because totality of data in development program showed that once daily 10-mg dapagliflozin provides optimal efficacy with safety and tolerance. Study continued to enroll with 2 arms.
Pre-assignment Details: 2245 enrolled. 1213 completed enrollment;1032 not completed:1 adverse event (AE), 65 withdrew consent (WC), 7 lost to follow up (LTF), 2 administrative (admin), 934 criteria not met, 2 non-compliant, 21 other. Lead-In: 588 randomized; 625 not randomized: 6 AE, 69 WC, 13 LTF, 8 admin, 2 at request, 497 criteria not met, 11 non-compliant, 19 other.
Groups:
- Placebo Matching Dapagliflozin: Placebo matching dapagliflozin: Tablets, Oral, 0 mg, once daily, Up to 12 weeks. Non-investigational medications used in this study were antidiabetic drug(s), including oral antidiabetic drugs and insulin, angiotensin-converting enzyme inhibitors or angiotensin receptor blockers, and an additional antihypertensive drug. All non-investigational medications were commercially available and were not supplied by the Sponsor.
- Dapagliflozin 10 mg: Dapagliflozin: Tablets, Oral, 10 mg, once daily, Up to 12 weeks. Non-investigational medications used in this study were antidiabetic drug(s), including oral antidiabetic drugs and insulin, angiotensin-converting enzyme inhibitors or angiotensin receptor blockers, and an additional antihypertensive drug. All non-investigational medications were commercially available and were not supplied by the Sponsor.
- Dagagliflozin 5 mg (Arm Discontinued With Amendment 8): Dapagliflozin: Tablets, Oral, 5 mg, once a day for up to12 weeks. Non-investigational medications used in this study were antidiabetic drug(s), including oral antidiabetic drugs and insulin, angiotensin-converting enzyme inhibitors or angiotensin receptor blockers, and an additional antihypertensive drug. All non-investigational medications were commercially available and were not supplied by the Sponsor.
  This arm was discontinued with Amendment 8 to the protocol (implemented 1 November 2011) and the other 2 arms continued to enroll. This arm is not included in primary and secondary efficacy analysis.
Period: Double Blind Treatment Period
Arm/Group | Placebo Matching Dapagliflozin | Dapagliflozin 10 mg | Dagagliflozin 5 mg (Arm Discontinued With Amendment 8)
Started | 224 | 225 | 133
Completed | 202 | 211 | 119
Not Completed | 22 | 14 | 14
Not completed — Adverse Event | 4 | 1 | 2
Not completed — Withdrawal by Subject | 6 | 4 | 4
Not completed — Lost to Follow-up | 3 | 2 | 3
Not completed — Administrative reason | 2 | 1 | 1
Not completed — Requested discontinue treatment | 1 | 0 | 1
Not completed — No Longer Meets Criteria | 1 | 5 | 2
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Non-specified | 3 | 0 | 0
Not completed — Missing disposition information | 0 | 1 | 1
Period: Follow-Up(Week 13/1 Week Post Last Dose)
Arm/Group | Placebo Matching Dapagliflozin | Dapagliflozin 10 mg | Dagagliflozin 5 mg (Arm Discontinued With Amendment 8)
Started | 203 (1 participant discontinued drug but remained in study and entered Follow-Up.) | 209 (2 participants completed treatment period but chose not to enter follow up period.) | 120 (1 participant discontinued drug but remained in the study and entered the follow up period.)
Completed | 200 | 209 | 119
Not Completed | 3 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — non-specified | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants in Double-Blind Period who were randomized and treated with at least one dose of double-blind study medication.
Groups:
- Dagagliflozin 5 mg (Arm Discontinued With Amendment 8): Dapagliflozin: Tablets, Oral, 5 mg, once daily, Up to 12 weeks. This arm discontinued with implementation of Amendment 8 to the protocol (1 November 2011). Study continued to enroll participants in other 2 arms post Amendment 8. Non-investigational medications used in this study were antidiabetic drug(s), including oral antidiabetic drugs and insulin, angiotensin-converting enzyme inhibitors or angiotensin receptor blockers, and an additional antihypertensive drug. All non-investigational medications were commercially available and were not supplied by the Sponsor.
- Total: Total of all reporting groups
Arm/Group | Placebo Matching Dapagliflozin | Dapagliflozin 10 mg | Dagagliflozin 5 mg (Arm Discontinued With Amendment 8) | Total
Number analyzed (Participants) | 224 | 225 | 133 | 582
Age, Customized [Number; unit: participants]
  Less than (<) 65 years | 198 | 198 | 118 | 514
  Greater than, equal (>=) to 65 and < 75 years | 25 | 23 | 14 | 62
  >= 75 years | 1 | 4 | 1 | 6
Gender [Count of Participants; unit: Participants]
  Female | 95 | 107 | 52 | 254
  Male | 129 | 118 | 81 | 328
Race/Ethnicity, Customized [Number; unit: participants] — Ethnicity was collected and summarized only for USA participants.
  participants
    White | 157 | 160 | 84 | 401
    Black or African American | 17 | 19 | 9 | 45
    Asian | 38 | 34 | 36 | 108
    Other Race | 12 | 12 | 4 | 28
    Ethnicity Hispanic/Latino | 41 | 47 | 21 | 109
    Ethnicity Not Hispanic/Latino | 40 | 38 | 16 | 94
    Ethnicity Not Reported | 143 | 140 | 96 | 379
Body Mass Index (BMI) [Number; unit: participants] — BMI is measured by weight in kilograms (kg) divided by height in meters (m) squared (kg/m^2). Less than (<); Greater than, equal to (>=).
  participants
    < 25 kg/m^2 | 21 | 17 | 9 | 47
    >=25 kg/m^2 | 203 | 208 | 124 | 535
    >=27 kg/m^2 | 179 | 178 | 101 | 458
    >=30 kg/m^2 | 147 | 141 | 73 | 361
Hypertension Medication [Number; unit: participants] — The following categories served as a randomization stratification factor:
  category 1: thiazide or thiazide-like diuretics and no insulin category 2: calcium channel blockers, beta blockers, central alpha adrenergic agonist or alpha adrenergic blockers and no insulin category 3: thiazide or thiazide-like diuretics and insulin category 4: calcium channel blockers, beta blockers, central alpha adrenergic agonist or alpha adrenergic blockers and insulin
  participants
    Thiazide or thiazide-like diuretics, no insulin | 94 | 95 | 54 | 243
    Calcium channel and beta blockers, no insulin | 114 | 112 | 79 | 305
    Thiazide or thiazide-like diuretics, insulin | 5 | 6 | 0 | 11
    Calcium channel and beta blockers, insulin | 11 | 12 | 0 | 23

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Seated Systolic Blood Pressure for 12 Week Double-Blind Treatment Period - Randomized Participants
Description: Systolic blood pressure (SBP) was measured in millimeters of mercury (mmHg) on Day -1, Day 1, Weeks 2, 4, 8, and 12 of the Double Blind Period. Blood pressure (BP) values were obtained after the participant was seated for quietly for 10 minutes; a mean of 3 replicate measurements was taken at least 1 minute apart. However, if the 3 consecutive seated BP readings were not within 8 mm Hg of each other, an additional 2 BP readings were obtained (total = 5) and incorporated into the calculated mean. BP was measured in both arms. If the BP was higher in one arm than the other, then this arm was used; if no difference, the participant's dominant arm was used for all future BP measurements. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. Participants refrained from ingestion of caffeine, alcohol, or nicotine at least 10 hours prior to their visit and having their BP measured.
Time Frame: Baseline to Week 12
Population: All randomized participants who received double-blind medication and had non-missing Baseline and on-study measurement. Data after rescue excluded from analyses
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo Matching Dapagliflozin | Dapagliflozin 10 mg
Number analyzed (Participants) | 218 | 221
mmHg
  Week 2 (N=218, 221) | -5.13 (0.9489) | -7.93 (0.9357)
  Week 4 (N=213, 220) | -6.05 (1.0232) | -9.69 (1.0097)
  Week 8 (N=205, 212) | -6.80 (1.0374) | -11.38 (1.0251)
  Week 12 (N=199, 205) | -7.62 (1.0701) | -11.90 (1.0585)
Statistical Analysis 1: Comparison: Placebo Matching Dapagliflozin vs Dapagliflozin 10 mg; Longitudinal repeated measures analysis using 'direct likelihood', with fixed categorical effects of treatment, week, treatment-by-week interaction, and randomization strata, as well as continuous fixed covariates of baseline SBP value and baseline SBP value-by-week interaction. Unstructured matrix for within-subject error variance-covariance used. 80% power to detect a difference of 4 mmHg in mean change from baseline, 75% power to meet both co-primary endpoints with overall Type I error; Test type: Superiority or Other; p = 0.0002, Longitudinal repeated measures — Endpoint was tested at alpha=0.05. Hierarchical closed testing procedure used; Data from all weeks during the double-blind treatment period were included; Mean Difference (Final Values) = -4.28, 95% CI 2-sided [-6.54 to -2.02], Standard Error of Mean 1.1485

2. Primary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1c (HbA1c) for 12 Week Double-Blind Treatment Period - Randomized Participants
Description: Adjusted mean change in glycosylated hemoglobin ( HbA1c) from baseline at Week 12 was calculated. HbA1c was measured as percent of hemoglobin by a central laboratory. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. HbA1c values were obtained at enrollment and lead-in (Day -28) periods, and at Day 1, Weeks 4, 8, and 12, in the double-blind period.
Time Frame: Baseline to Week 12
Population: All randomized participants who received double-blind medication and had non-missing Baseline and on-study measurement. Data after rescue included.
Measure: Mean (Standard Error); unit: Percent of Hemoglobin
Arm/Group | Placebo Matching Dapagliflozin | Dapagliflozin 10 mg
Number analyzed (Participants) | 214 | 219
Percent of Hemoglobin
  Week 4 (N=214, 219) | -0.06 (0.0498) | -0.41 (0.0496)
  Week 8 (N=207, 211) | -0.07 (0.0606) | -0.58 (0.0602)
  Week 12 (N=197, 204) | -0.02 (0.0673) | -0.63 (0.0668)
Statistical Analysis 1: Comparison: Placebo Matching Dapagliflozin vs Dapagliflozin 10 mg; A longitudinal repeated measures analysis used, with fixed categorical effects of treatment, week, treatment-by-week interaction, and randomization strata, continuous fixed covariates of baseline HbA1c value and baseline HbA1c value-by-week interaction. Only data up to Week 12 included. All data used in the model even if participants discontinued prior to Week 12. A heirarchical closed testing procedure (sequential) was used and testing performed since first primary endpoint was significant; Test type: Superiority or Other; p < 0.0001, Longitudinal repeated measures; Endpoint was tested at alpha=0.05. Hierarchical closed testing procedure was used; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.76 to -0.46], Standard Error of Mean 0.0773

3. Secondary Outcome: Adjusted Mean Change From Baseline in 24-hour Ambulatory Systolic Blood Pressure at Week 12 Last Observation Carried Forward (LOCF)
Description: Ambulatory 24 hour (hr) blood pressure monitoring (ABPM) was performed at baseline, which was during the lead-in period (between Day -7 and Day -1 prior to randomization) and 1 week prior to the Week 12 visit/end of treatment visit. If no Week 12 measurement was available, the last available earlier post-baseline measurement was used (LOCF) for analysis. Initiation of the 24-hr ABPM began between 6am and 11am to ensure trough BP measurements were obtained.The ABPM units were calibrated, and used per the manufacturer's and central ABPM vendor instructions. BP was measured in mmHg. Participants had to have a mean 24-hour ABPM ≥ 130/80 mmHg prior to randomization. All medication was withheld on the morning of the study visit and brought to the visit site by the participant. Once the ABPM cuff was in place, all morning medication was taken while at the site.
Time Frame: Baseline, Week 12
Population: All randomized participants who received double-blind medication and had non-missing Baseline and Week 12 (LOCF) values. Data after rescue excluded from analyses.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo Matching Dapagliflozin | Dapagliflozin 10 mg
Number analyzed (Participants) | 186 | 187
mmHg | -6.88 (1.5793) | -11.33 (1.6031)
Statistical Analysis 1: Comparison: Placebo Matching Dapagliflozin vs Dapagliflozin 10 mg; ANCOVA model with treatment group as an effect and baseline value and randomization strata as a covariate was used. By applying sequential testing procedure, the testing was performed since the prior endpoint was significant; Test type: Superiority or Other; p = 0.0012, ANCOVA — Endpoint tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -4.45, 95% CI 2-sided [-7.14 to -1.76], Standard Error of Mean 1.3680

4. Secondary Outcome: Adjusted Mean Change From Baseline in Seated Diastolic Blood Pressure (DBP) for 12 Week Double-Blind Treatment Period - Randomized Participants
Description: Diastolic BP was measured in millimeters of mercury (mmHg) on Day -1, Day 1, Weeks 2, 4, 8, and 12 of the Double Blind Period. Diastolic BP values were obtained after the participant was seated for quietly for 10 minutes; a mean of 3 replicate measurements was taken at least 1 minute apart. However, if the 3 consecutive seated BP readings were not within 8 mm Hg of each other, an additional 2 BP readings were obtained (total = 5) and incorporated into the calculated mean. BP was measured in both arms. If the pressure was higher in one arm than the other, then this arm was used; if no difference, the participant's dominant arm was used for all future BP measurements. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. Participants refrained from ingestion of caffeine, alcohol, or nicotine at least 10 hours prior to their visit and having their BP measured.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Placebo Matching Dapagliflozin: Placebo matching dapagliflozin: Tablets, Oral, 0 mg, once daily, Up to 12 weeks.Non-investigational medications used in this study were antidiabetic drug(s), including oral antidiabetic drugs and insulin, angiotensin-converting enzyme inhibitors or angiotensin receptor blockers, and an additional antihypertensive drug. All non-investigational medications were commercially available and were not supplied by the Sponsor.
Arm/Group | Placebo Matching Dapagliflozin | Dapagliflozin 10 mg
Number analyzed (Participants) | 218 | 221
mmHg
  Week 2 (N=218, 221) | -3.84 (0.5691) | -5.22 (0.5613)
  Week 4 (N=213, 220) | -4.28 (0.5894) | -5.57 (0.5818)
  Week 8 (N=205, 212) | -4.76 (0.6247) | -6.53 (0.6170)
  Week 12 (N=199, 205) | -5.33 (0.6377) | -6.30 (0.6308)
Statistical Analysis 1: Comparison: Placebo Matching Dapagliflozin vs Dapagliflozin 10 mg; Longitudinal repeated measures analysis using direct likelihood with fixed categorical effects of treatment, week, treatment-by week interaction, and randomization strata and continuous fixed covariates of baseline seated diastolic BP value and baseline seated diastolic BP value by week interaction; Test type: Superiority or Other; p = 0.1619, Longitudinal repeated measures — Endpoint tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-2.32 to 0.39], Standard Error of Mean 0.6900

5. Secondary Outcome: Adjusted Mean Change From Baseline in 24-hr Ambulatory Diastolic Blood Pressure at Week 12 (LOCF)
Description: Ambulatory 24 hour (hr) BP monitoring (ABPM) was performed at baseline, which was during the lead-in period (between Day -7 and Day -1 prior to randomization) and 1 week prior to the Week 12 visit/end of treatment visit. If no Week 12 measurement was available, the last available earlier post-baseline measurement was used (LOCF). Initiation of the 24-hr ABPM began between 6am and 11am to ensure trough BP measurements were obtained. The ABPM units were calibrated, and used per the manufacturer's and central ABPM vendor instructions. BP was measured in mmHg. Participants had to have a mean 24-hour ABPM ≥ 130/80 mmHg prior to randomization. All medication was withheld on the morning of the study visit and brought to the visit site by the participant. Once the ABPM cuff was in place, all morning medication was taken while at the site.
Time Frame: Baseline, Week 12
Population: All randomized participants who received double-blind medication and had non-missing Baseline and on-study measurement (Week 12 LOCF). Data after rescue excluded from analyses.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo Matching Dapagliflozin | Dapagliflozin 10 mg
Number analyzed (Participants) | 186 | 187
mmHg | -5.57 (1.0042) | -7.56 (1.0183)
Statistical Analysis 1: Comparison: Placebo Matching Dapagliflozin vs Dapagliflozin 10 mg; ANCOVA model with treatment group as an effect and baseline value and randomization strata as a covariate. A hierarchical closed testing procedure was implemented to control the family-wise type I error rate related to the co-primary and secondary endpoints at the 2-sided 0.05 level. Statistical testing of this endpoint was not performed since the prior secondary endpoint was not statistically significant; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.99, 95% CI 2-sided [-3.68 to -0.29], Standard Error of Mean 0.8635

6. Secondary Outcome: Adjusted Mean Change From Baseline in Serum Uric Acid at Week 12 in Double-Blind Treatment Period - Randomized Participants
Description: Adjusted mean change in serum uric acid from baseline at Week 12 was calculated. Serum uric acid was measured in milligrams per deciliter (mg/dL) by a central laboratory. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. Serum uric acid measurements were obtained at qualification and lead-in (Day -28) periods, and at Day 1, Weeks 4, 8, and 12, in the double-blind period but only the change from baseline at Week 12 was considered a secondary endpoint and is presented.
Time Frame: Baseline, Week 12
Population: All randomized participants who received double-blind medication and had non-missing Baseline and on-study measurement. Data after rescue was included.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo Matching Dapagliflozin | Dapagliflozin 10 mg
Number analyzed (Participants) | 210 | 219
mg/dL | -0.03 (0.0890) | -0.43 (0.0883)
Statistical Analysis 1: Comparison: Placebo Matching Dapagliflozin vs Dapagliflozin 10 mg; Longitudinal repeated measures analysis using direct likelihood with fixed categorical effects of treatment, week, treatment-by week interaction, and randomization strata and continuous fixed covariates of baseline serum uric acid value and baseline seated serum uric acid value by week interaction. By applying sequential testing procedure at alpha=0.05, no testing was performed since the prior secondary endpoint was not significant; Test type: Superiority or Other; lLongitudinal repeated measures; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.57 to -0.23], Standard Error of Mean 0.0858

7. Secondary Outcome: Number of Participants With Deaths,Serious Adverse Events (SAEs), Adverse Events (AEs), Hypoglycemia Events, Discontinuation Due to AEs, SAEs and Hypoglycemia, During the 12 Week Double Blind Period, Including Data After Rescue
Description: Medical Dictionary for Regulatory Activities (MedDRA), version 15.1 AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Related=having certain, probable, possible, or missing relationship to study drug as per the investigator. Events captured from baseline to last double blind dose plus 4 days for AEs, plus 30 days for SAEs during the Double Blind 12 Week Period. Only hypoglycemia reported as an SAE is included in AE/SAE categories . All reported hypoglycemia events within 4 days of last day of treatment are included as hypoglycemic events.
Time Frame: Baseline to last dose of 12 weeks of double blind medication plus 30 days if SAE or plus 4 days if AE/hypoglycemic event
Population: Randomized participants who received double-blind study medication in the double-blind period.
Measure: Number; unit: participants
Arm/Group | Placebo Matching Dapagliflozin | Dapagliflozin 10 mg | Dagagliflozin 5 mg (Arm Discontinued With Amendment 8)
Number analyzed (Participants) | 224 | 225 | 133
participants
  Deaths | 0 | 0 | 0
  SAEs | 2 | 6 | 1
  Related SAEs | 1 | 0 | 0
  AEs | 93 | 98 | 60
  Hypoglycemia AEs | 6 | 13 | 2
  Related AEs | 12 | 15 | 8
  Discontinued due to AE | 4 | 1 | 2
  Discontinued due to SAE | 1 | 0 | 1
  Discontinued due to Hypoglycemia | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Marked Chemistry Laboratory Abnormalities in 12 Week Double Blind Treatment Period, Including Data After Rescue
Description: Samples obtained: Day 1, Weeks 4, 8,12 in Double Blind Period. Baseline: last assessment prior to start of first dose of double-blind treatment. Pretreatment (PreRX); grams per deciliter (g/dL); upper limit of normal (ULN); milliequivalent per liter (mEq/L); greater than (>) less than (<); Units per liter (U/L), Marked abnormality Low (High): hemoglobin <6 (>18 females or >20 males) g/dL; creatinine (>=1.5*preRX, >=2.5 mg/dL); glucose < 54 or (> 350) mg/dL; albumin <= 2 or (> 6) g/dL; creatine kinase >5*ULN; albumin/creatinine ratio (>1800 mg/G); calcium <7.5 (>1 and >0.5 from PreRX) mg/dL; bicarbonate <=13 meq/dL; potassium <=2.5 (>6) meq/L; magnesium <1 (>4) mEq/L; sodium < 130 mEq/L (>150 mEq/L; phosphorus (>=5.6 mg/dL age 17-65, >=5.1 is >=66 years); Albumin/creatinine ratio (>1800 mg/g). Note: Hepatic tests are presented separately in next outcome measure.
Time Frame: Baseline (Day 1) to last dose double blind medication (Week 12) plus 4 days
Population: N=All randomized participants who received at least one dose of double-blind medication. n=all treated participants who had non-missing Baseline and on-study measurement. Data after rescue included.
Measure: Number; unit: participants
Arm/Group | Placebo Matching Dapagliflozin | Dapagliflozin 10 mg
Number analyzed (Participants) | 218 | 223
participants
  Hemoglobin High >18 g/dL (n=218, 223) | 1 | 0
  Creatinine >=1.5PreRx (n=218,223) | 1 | 3
  Glucose, plasma unspecif <54 mg/dL (n=218,222) | 0 | 1
  Glucose, plasma unspecif >350 mg/dL (n=218,222) | 2 | 1
  Creatine Kinase >5*ULN (n=218,223) | 2 | 0
  Creatine Kinase >10*ULN (n=218,223) | 1 | 0
  Calcium, total <7.5 mg (n=218,223) | 0 | 1
  Potassium, serum≥6 mEq/L (n=218,222) | 0 | 4
  Magnesium <1 mEq/L (n=218,223) | 0 | 2
  Sodium, serum <130 mEq/L (n=218,222) | 1 | 0
  Sodium, serum >150 mEq/L (n=218,222) | 1 | 1
  Phosphorus inorganic High (n=218,223) | 0 | 2
  Albumin/Creatinine Ratio High (n=218, 223) | 5 | 3

9. Secondary Outcome: Number of Participants With Elevated Liver Laboratory Tests in Participants Treated With Double Blind 10 mg Dapagliflozin or Placebo , Including Data After Rescue
Description: Laboratories were obtained at Day 1, Weeks 4, 8 and 12 in the Double Blind Period. Baseline: last assessment prior to start of first dose of double-blind treatment. Includes laboratory values measured after the first date of double-blind treatment and up to and including the last day of double blind treatment plus 30 days. Upper limit of normal (ULN);, alanine aminotransferase (ALT); aspartate aminotransferase (AST); alkaline phosphatase (ALP). Marked abnormality (High): AST and ALT (>3*ULN); ALP (>1.5*ULN); bilirubin (>1.5*ULN). Participants with abnormally elevated liver laboratory tests were followed 30 days after the last dose of study drug.
Time Frame: Baseline (Day 1) to last dose double blind medication (Week 12) Plus 30 days
Population: N=All randomized participants who received at least 1 dose of study medication. n=number of participants treated with double blind study medication with at least one non-missing post-baseline value. Data after rescue included.
Measure: Number; unit: participants
Arm/Group | Placebo Matching Dapagliflozin | Dapagliflozin 10 mg
Number analyzed (Participants) | 221 | 224
participants
  AST >3*ULN (n=221, 224) | 0 | 3
  AST >5*ULN (n=221, 224) | 0 | 1
  AST >10*ULN (n=221, 224) | 0 | 1
  AST >20*ULN (n=221, 224) | 0 | 1
  ALT >3*ULN (n=221, 224) | 0 | 3
  ALT >5*ULN (n=221, 224) | 0 | 2
  ALT >10*ULN (n=221, 224) | 0 | 1
  ALT >20*ULN (n=221, 224) | 0 | 1
  Total Bilirubin >1.5*ULN (n=221, 224) | 0 | 2
  Total Bilirubin >2*ULN (n=221, 224) | 0 | 1
  ALP >1.5*ULN (n=221, 224) | 5 | 4

10. Secondary Outcome: Number of Participants With Normal or Abnormal Electrocardiogram Summary Tracing at Week 12 (LOCF), Including Data After Rescue
Description: 12-Lead electrocardiograms (ECGs) were performed at Enrollment, Day 1 of Double Blind Period and Week 12/End of treatment visit (last observation carried forward) on participants who were supine. ECGs were assessed by the investigator as normal or abnormal. Baseline (BL) was Day 1 prior to dosing or last observation prior to dosing.
Time Frame: Baseline, Week 12
Population: N= All randomized participants who received double-blind medication. Data after rescue included.
Measure: Number; unit: participants
Arm/Group | Placebo Matching Dapagliflozin | Dapagliflozin 10 mg
Number analyzed (Participants) | 224 | 225
participants
  Baseline normal/Week 12 normal | 137 | 130
  Baseline normal/Week 12 abnormal | 9 | 10
  Baseline normal/ Week 12 not reported | 0 | 0
  Baseline abnormal/Week 12 normal | 10 | 22
  Baselline abnormal/Week 12 abnormal | 48 | 50
  Baseline abnormal/Week 12 not reported | 0 | 0
  Baseline not reported/Week 12 normal | 0 | 0
  Baseline not reported/Week 12 abnormal | 0 | 0
  Baseline not reported/Week 12 not reported | 20 | 13

11. Secondary Outcome: Proportion of Participants With Orthostatic Hypotension at Baseline and Week 12, Including Data After Rescue
Description: Orthostatic hypotension was defined as a decrease from supine to standing of > 20 mmHg in systolic BP or >10 mmHg in diastolic BP. Proportion was calculated from number of participants with orthostatic hypotension (n) divided by the number of treated participants (N). n/N presented as a percent (%). Baseline was Day 1 of the double blind Period. Measurements for orthostatic hypotension were taken on Day 1 and at Week 12 visit and does not reflect AEs reported by the investigator.
Time Frame: Baseline (Day 1), Week 12
Population: N= All randomized participants who received double-blind medication and had non-missing Week (t) values. Week 12 includes participants with orthostatic hypotension during Week 12 visit window. Data after rescue included.
Measure: Number; unit: Percent of Participants
Arm/Group | Placebo Matching Dapagliflozin | Dapagliflozin 10 mg
Number analyzed (Participants) | 220 | 222
Percent of Participants
  Baseline n/N (2/220, 2/222) | 0.9 | 0.9
  Week 12 n/N (4/199, 7/203) | 2.0 | 3.4

ADVERSE EVENTS:
Time Frame: 12 Weeks plus 30 days
Description: Baseline to last dose of 12 weeks of double blind medication plus 30 days if SAE or plus 4 days if AE/hypoglycemic event
Arm/Group | Placebo Matching Dapagliflozin | Dapagliflozin 10 mg | Dagagliflozin 5 mg (Arm Discontinued With Amendment 8)
Serious Adverse Events (participants affected / at risk) | 2/224 | 6/225 | 1/133
Other Adverse Events (participants affected / at risk) | 0/224 | 0/225 | 0/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching Dapagliflozin (N=224) | Dapagliflozin 10 mg (N=225) | Dagagliflozin 5 mg (Arm Discontinued With Amendment 8) (N=133)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hepatitis E (Infections and infestations) | 0 | 1 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Totality of data from dapagliflozin development program as of 1 NOV 2011 showed 10 mg dapagliflozin dose provided optimal efficacy, was safe and well tolerated for the general Type 2 diabetes population, allowing the 5 mg arm to be discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.